CLINICAL TRIAL: NCT01034384
Title: Physiological, Cognitive and Cerebral Activity Changes as a Function of Cigarette Smoking (With or Without Nicotine) and Tobacco Abstinence
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901357; 01-DA-N357
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2012-11-06

CONDITIONS: Smoking Cessation
Keywords: fMRI; Smoking Withdrawal; Imaging; Memory; Mood
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Denicotinized cigarettes are similar to commercial cigarettes but contain and deliver virtually no nicotine. Denicotinized cigarettes are used as a control condition in smoking research, as a substitute treatment for nicotine dependence, and as a strategy to reduce incidence of nicotine addiction. However, the symptoms of nicotine withdrawal and craving for cigarettes must be minimized to ensure that smokers will continue to use denicotinized cigarettes instead of their preferred cigarettes.
* Although research has shown that smokers preferred cigarettes that delivered nicotine, subjective measures of tobacco craving and withdrawal were similar after standard and denicotinized cigarettes. This suggests that the process of smoking and non-nicotine components of tobacco smoke mediate some of the effects of cigarette smoking. More research is needed on the comparative physical and mental effects of regular cigarettes and denicotinized cigarettes.

Objectives:

- To compare the effects of complete abstinence or smoking denicotinized cigarettes with smoking nicotinized cigarettes on the following measures: (1) withdrawal symptoms and quality of sleep, (2) hormonal responses, (3) mood and cognitive performance, and (4) functional brain activity.

Eligibility:

- Men between 18 and 50 years of age who are either current smokers (at least 15 cigarettes per day for at least 2 years) or nonsmoking volunteers.

Design:

* Participants will be divided into four groups: (1) nonsmokers, (2) smokers who receive nicotinized cigarettes, (3) smokers who receive denicotinized cigarettes, and (4) smokers who will abstain from cigarettes.
* The study will last 16 days. Smokers will have 14 visits to the clinical center; nonsmokers will have 6 visits. From Day 6 to Day 14, current smokers will follow the smoking regimen assigned by the researchers (not smoking, smoking denicotinized cigarettes, or smoking nicotinized cigarettes).
* Nonsmokers will have one day of training on the memory and thinking tasks that will be performed in the functional magnetic resonance imaging (fMRI) scanner, and will have 5 additional days of two fMRI scans per day (total of 10 fMRI scans).
* Current smokers will have 2 days of training on the memory and thinking tasks that will be performed in the fMRI scanner, physical assessments on Day 3 and Day 6, and 5 days of two fMRI scans per day (total of 10 fMRI scans).
* Participants in the complete abstinence group will be asked to resume smoking after the abstinence period and the denicotinized cigarettes group will resume nicotinized cigarettes on day 14. Participants can decline to resume smoking, and if desired they will be referred for smoking cessation treatment.

DETAILED DESCRIPTION:
Objective:

To compare the effects of complete abstinence or smoking denicotinized research cigarettes to smoking ad libitum nicotinized research cigarettes on the following measures: withdrawal symptoms and quality of sleep; MAO-A and MAO-B activities; hormonal responses (HPA, HPT); mood, cognitive and psychometric performance; functional brain activity, and physiological responses.

Study Population:

Participants are 125 men who are at least 18 years old, report smoking at least 15 cigarettes per day, have not used any illicit drug except marijuana in the past year, have no history of drug or alcohol dependence, and have already experienced tobacco withdrawal symptoms when they had no access to cigarettes.

Design:

Smokers will be randomized into one of the following 3 groups: a) complete tobacco abstinence for 8 days; b) denicotinized research cigarettes for 8 days, or c) control group smoking nicotinized research cigarettes during the entire study (16 days). Because there are few studies comparing functional brain activity in smokers and nonsmokers, a group of nonsmokers will serve as a control group for the brain imaging studies.

Outcome Measures:

Withdrawal symptoms, mood, quality of sleep, cognitive performance, temperature, blood pressure and heart rate, MAO-A parameters: plasma DHPG (dihydroxyphenylglycol), HVA (homovanillic acid), 5HIAA (5-hydroxyindolacetic acid); MAO-B parameters: urinary excretion of phenylethylamine, platelet MAO-B activity; hormonal parameters: serum ACTH, cortisol, TSH, thyroxine, triiodothyronine; EEG; cigarette liking; expired air CO; and functional brain activity.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must be:

1. Between the ages of 18-50.
2. In good health.
3. Right-handed.
4. Free of past or present abuse and dependence on other substances (except nicotine).
5. Able to abstain from alcohol for 24 hours before each experiment session and no more than 50 mg of caffeine (about 1/2 cup of coffee or a 12 oz cola) for 12 hours before each neuroimaging session.
6. Male.

Smokers must be:

1. Regular smokers of greater than or equal to 15 cigarettes other than ultra-low nicotine cigarettes per day for at least two years with evidence of withdrawal symptoms when having stopped smoking for several hours (planes, theater, etc).

Nonsmokers must:

1. Have smoked less than or equal to 5 cigarettes in their lifetime, and no cigarettes or any tobacco product in the past 5 years, and expired air CO < 8ppm.

EXCLUSION CRITERIA:

Participants will be excluded if they:

1. Are not suitable to undergo an fMRI experiment due to implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology or claustrophobia.
2. Have coagulopathies, history of or current superficial, or deep vein thrombosis, or musculoskeletal abnormalities restricting an individual s ability to lie flat for extended periods of time.
3. Have HIV or Syphilis.
4. Have any neurological illnesses to include, but not limited to, seizure disorders, migraine (>2/yr or on prophylaxis), multiple sclerosis, movement disorders, or history of significant head trauma, CVA, CNS tumor.
5. Have other major medical illnesses likely to interfere with study results or safety of an individual during participation.

   * Hemoglobin < 10 g/dl
   * White Blood Cell Count < 2400/microliters
   * Liver Function Tests > 3 times normal
   * Serum glucose > 200 mg/dl
   * Urine protein > 2 plus
6. Have any current major psychiatric disorders to include, but not limited to, mood, anxiety, psychotic disorders, or substance-induced psychiatric disorders.
7. Regularly use any prescription, over-the-counter or herbal medication that may alter CNS function, cardiovascular function or neuronal-vascular coupling.
8. Are cognitively impaired or learning disabled.
9. Significant cardiovascular or cerebrovascular diseases.

INCLUSION CRITERIA (Pilot Studies):

Smokers:

* regular cigarette smokers smoking greater than or equal to 10 cigarettes/day for at least 1 year
* no intention to reduce or quit tobacco use
* age between 18 and 45 years
* men

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2000-12-05; Study Completion 2012-11-06

PRIMARY OUTCOMES:
Subjective withdrawal symptoms, cognitive performance, vital signs, MAO-A and MAO-B parameters, hormonal parameters, EEG, cigarette liking, expired air CO, and functional brain activity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Heishman, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States